CLINICAL TRIAL: NCT01892020
Title: A Multi-centre, Randomised, Open-labelled, 2-sequence, 2-period Crossover Trial to Investigate the Efficacy and Safety of Biphasic Insulin Aspart 50 (BIAsp 50) Twice Daily Versus Biphasic Human Insulin 50 (BHI 50) Twice Daily Both in Combination With Metformin in Chinese Subjects With Type 2 Diabetes Mellitus
Brief Title: Investigating Efficacy and Safety of Biphasic Insulin Aspart 50 Twice Daily Versus Biphasic Human Insulin 50 Twice Daily Both in Combination With Metformin in Chinese Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-4058; U1111-1137-2342 (Other: WHO)
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence 1 (Group A) (Experimental): Group A will receive BIAsp 50 BID during the first 4 weeks (treatment period 1) then switch to BHI 50 BID for further 4 weeks (treatment period 2)
  Interventions: Drug: biphasic insulin aspart 50; Drug: biphasic human insulin 50
- Treatment sequence 2 (Group B) (Experimental): Group B will receive BHI 50 BID during the first 4 weeks (treatment period 1), then switch to BIAsp 50 BID for further 4 weeks (treatment period 2)
  Interventions: Drug: biphasic insulin aspart 50; Drug: biphasic human insulin 50

INTERVENTIONS:
Drug: biphasic insulin aspart 50 — Administered subcutaneously (s.c., under the skin) twice daily (BID). Dose individually adjusted. All subjects will receive metformin in combination with trial insulin.
Drug: biphasic human insulin 50 — Administered subcutaneously (s.c., under the skin) twice daily (BID). Dose individually adjusted. All subjects will receive metformin in combination with trial insulin.

SUMMARY:
This trial is conducted in Asia. The aim of the trial is to investigate the efficacy and safety of biphasic insulin aspart 50 (BIAsp 50) twice daily versus biphasic human insulin 50 (BHI 50) twice daily, both in combination with metformin, in Chinese subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (diagnosed clinically) for at least 12 months
* Currently treated with premixed human insulin 50 BID for at least 3 months prior to screening visit (Visit 1)
* Currently treated with unchanged total daily dose of at least 1500 mg metformin or maximum tolerated dose at least 1000 mg/day metformin for at least 2 months prior to screening visit
* Glycosylated haemoglobin (HbA1c) 7.0% and 9.0% (both inclusive) (central laboratory)

Exclusion Criteria:

* Treatment with any insulin secretagogue, alfa-glucosidase inhibitors, thiazolidinedione (TZD), dipeptidyl peptidase-4 (DPP-4) inhibitors and Glucagon-like peptide-1 (GLP-1) receptor agonists within the last 3 months prior to screening
* Previous use of any insulin other than premixed human insulin 50 BID within 3 months prior to Visit 1
* Previous use of insulin intensification treatment (premixed insulin thrice daily, basal bolus regimen, and continuous subcutaneous insulin infusion (CSII)) for more than 14 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Beijing, Beijing Municipality, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 14 sites in one country (China).
Pre-assignment Details: There were no significant events following enrolment of subjects, and prior to randomization.
Groups:
- Group A (BIAsp 50 - BHI 50): In this multi-center, randomized, open-labelled, 2-sequence, 2-period crossover trial, the eligible subjects were randomized to 2 groups to receive biphasic insulin aspart 50 (BIAsp 50) and biphasic human insulin 50 (BHI 50) in different sequences.
  Group A received BIAsp 50 twice daily (BID) during the first 4 weeks (period 1), then switched to BHI 50 BID for further 4 weeks (period 2). BIAsp 50 (NovoMix® 50) was administered subcutaneously (s.c.) using NovoPen 4 immediately before breakfast and dinner. And BHI 50 was administered s.c. using NovoPen 4 at least 30 minutes before breakfast and dinner. All subjects received metformin throughout this trial. Insulin dose was adjusted twice weekly based on self-measured plasma glucose (SMPG).
- Group B (BHI 50 - BIAsp 50): In this multi-center, randomized, open-labelled, 2-sequence, 2-period crossover trial, the eligible subjects were randomized to 2 groups to receive biphasic insulin aspart 50 (BIAsp 50) and biphasic human insulin 50 (BHI 50) in different sequences.
  Group B received BHI 50 twice daily (BID) during the first 4 weeks (period 1), then switched to BIAsp 50 BID for further 4 weeks (period 2). BIAsp 50 (NovoMix® 50) was administered subcutaneously (s.c.) using NovoPen 4 immediately before breakfast and dinner. And BHI 50 was administered s.c. using NovoPen 4 at least 30 minutes before breakfast and dinner. All subjects received metformin throughout this trial. Insulin dose was adjusted twice weekly based on self-measured plasma glucose (SMPG).
Period: Period 1
Arm/Group | Group A (BIAsp 50 - BHI 50) | Group B (BHI 50 - BIAsp 50)
Started | 81 | 80
Completed | 78 | 74
Not Completed | 3 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 2 | 4
Not completed — Unclassified | 0 | 1
Period: Period 2
Arm/Group | Group A (BIAsp 50 - BHI 50) | Group B (BHI 50 - BIAsp 50)
Started | 78 | 74
Completed | 77 | 74
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: In this multi-center, randomized, open-labelled, 2-sequence, 2-period crossover trial, the eligible subjects were randomized to 2 groups to receive biphasic insulin aspart 50 (BIAsp 50) and biphasic human insulin 50 (BHI 50) in different sequences. Group A received BIAsp 50 twice daily (BID) during the first 4 weeks (period 1), then switched to BHI 50 BID for further 4 weeks (period 2). Group B received BHI 50 BID during the first 4 weeks (period 1), then switched to BIAsp 50 BID for further 4 weeks (period 2). BIAsp 50 (NovoMix® 50) was administered subcutaneously (s.c.) using NovoPen 4 immediately before breakfast and dinner. And BHI 50 was administered s.c. using NovoPen 4 at least 30 minutes before breakfast and dinner. All subjects received metformin throughout this trial. Insulin dose was adjusted twice weekly based on self-measured plasma glucose (SMPG).
Arm/Group | All Subjects
Number analyzed (Participants) | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 73

OUTCOME MEASURES:

1. Primary Outcome: 2-hour PPG (Postprandial Plasma Glucose) Increment Following a Standard Meal Test
Description: The 2-hour PPG increment is the difference between the plasma glucose (PG) value at 120 minutes after standard meal test and the fasting PG value.
Time Frame: After 4 weeks of treatment in each treatment sequence
Population: Of the 161 randomized subjects, 155 subjects received BIAsp 50 and 158 subjects received BHI 50 (152 subjects received both, 3 subjects only received BIAsp 50 and 6 subjects only received BHI 50). Three (3) subjects in BIAsp 50 group and 9 subjects in BHI 50 group did not contribute to the analysis due to lack of post-randomization measurements.
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- BIAsp 50: This arm included the subjects received BIAsp 50.
- BHI 50: This arm included the subjects received BHI 50.
Arm/Group | BIAsp 50 | BHI 50
Number analyzed (Participants) | 152 | 149
mmol/L | 5.30 (3.17) | 6.41 (2.83)
Statistical Analysis 1: Comparison: BIAsp 50 vs BHI 50; Let D be the treatment difference (BIAsp 50 BID + metformin minus BHI 50 BID + metformin) of 2-h PPG increment after a 4-week treatment. The null hypothesis was D = 0 mmol/L. The alternative hypothesis was D ≠ 0 mmol/L. Sample size was determined using a two-sided one sample t-test at a = 0.05 under the assumption of 0.8 mmol/L mean treatment different and 80% power; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The 2-h PPG increment was analyzed using a normal linear mixed model with period and treatment as fixed effects and subject as a random effect; Mean Difference (Net) = -1.12, 95% CI [-1.66 to -0.58], Standard Error of Mean 0.27

2. Secondary Outcome: -1-hour PPG Increment Following a Standard Meal Test
Description: The 1-h PPG increment is the difference between the plasma glucose (PG) value at 60 minutes after standard meal test and the fasting PG value.
Time Frame: After 4 weeks of treatment in each treatment sequence
Population: Of the 161 randomized subjects, 155 subjects received BIAsp 50 and 158 subjects received BHI 50 (152 subjects received both, 3 subjects only received BIAsp 50 and 6 subjects only received BHI 50). Three (3) subjects in BIAsp 50 group and 8 subjects in BHI 50 group did not contribute to the analysis due to lack of post-randomization measurements.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | BIAsp 50 | BHI 50
Number analyzed (Participants) | 152 | 150
mmol/L | 4.42 (2.49) | 4.74 (2.24)

3. Secondary Outcome: -IAUC (Incremental Area Under the Curve) for PPG (0-2 Hours) Following a Standard Meal Test
Description: AUC for plasma glucose was calculated by the trapezoidal method using 30-min sampling time points, and IAUC for PPG (0-2h) data was analyzed using a normal linear mixed model.
Time Frame: After 4 weeks of treatment in each treatment sequence
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: min*mmol/L
Arm/Group | BIAsp 50 | BHI 50
Number analyzed (Participants) | 152 | 149
min*mmol/L | 465.39 (228) | 503.64 (215)

4. Secondary Outcome: 2-hour PPG Increments Over Each of the 3 Main Meals in 8-point SMPG (Self-measured Plasma Glucose) Profile
Description: PPG increments over each of the 3 main meals were derived from the 8-point SMPG profile as the difference between PG values available 120 minutes after meal and before meal.
Time Frame: After 4 weeks of treatment in each treatment sequence
Population: Of the 161 randomized subjects, 155 subjects received BIAsp 50 and 158 subjects received BHI 50 (152 subjects received both, 3 subjects only received BIAsp 50 and 6 subjects only received BHI 50). Subjects were excluded from analysis due to lack of post-randomization measurements. See table.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BIAsp 50 | BHI 50
Number analyzed (Participants) | 151 | 149
mmol/L
  Increment at breakfast, N=151, 149 | 2.52 (0.20) | 2.86 (0.20)
  Increment at Lunch, N=150, 148 | 3.58 (0.26) | 2.93 (0.26)
  Increment at dinner, N=151, 149 | 1.08 (0.26) | 0.99 (0.26)

5. Secondary Outcome: The Mean 2-hour PPG Increments of the 3 Main Meals in 8-point SMPG Profile
Description: Mean post prandial PG increment over all meals was derived as the mean of all available meal increments.
Time Frame: After 4 weeks of treatment in each treatment sequence
Population: Of the 161 randomized subjects, 155 subjects received BIAsp 50 and 158 subjects received BHI 50 (152 subjects received both, 3 subjects only received BIAsp 50 and 6 subjects only received BHI 50). Four (4) subjects in BIAsp 50 group and 9 subjects in BHI 50 group did not contribute to the analysis due to lack of post-randomization measurements.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BIAsp 50 | BHI 50
Number analyzed (Participants) | 151 | 149
mmol/L | 2.39 (0.15) | 2.25 (0.15)

6. Secondary Outcome: Incidence of Hypoglycemic Episodes
Description: Treatment Emergent Hypoglycemic Episode refers to those the onset of the episode is on or after the first day of exposure to randomized treatment and no later than the last day of randomized treatment. Results are presented by American Diabetes Association classification of hypoglycemia.
Time Frame: During 4 weeks of treatment in each treatment sequence
Population: Safety analysis set included all subjects receiving at least one dose of investigational products.
Measure: Number; unit: events per patient per year
Arm/Group | BIAsp 50 | BHI 50
Number analyzed (Participants) | 155 | 158
events per patient per year
  All events | 12.10 | 14.38
  Severe | 0 | 0.08
  Documented Symptomatic | 5.97 | 8.33
  Asymptomatic | 1.29 | 2.53
  Probable Symptomatic | 2.58 | 1.72
  Relative | 2.10 | 1.72
  Unclassifiable | 0.16 | 0

7. Secondary Outcome: Incidence of AEs (Adverse Event)
Description: Treatment emergent AE (TEAE) is defined as an event that has onset date on or after the first day of exposure to randomized treatment and no later than the last day of randomized treatment.
Time Frame: During 4 weeks of treatment in each treatment sequence
Population: Safety analysis set included all subjects receiving at least one dose of investigational products.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | BIAsp 50 | BHI 50
Number analyzed (Participants) | 155 | 158
Events/100 years of patient exposure | 322.7 | 245.1

ADVERSE EVENTS:
Time Frame: An event with onset date on or after the first day of exposure to randomized treatment and no later than the last day of randomized treatment was defined as treatment emergent AE. All events meeting this definition were collected and reported.
Description: Safety analysis set included all subjects receiving at least one dose of investigational products.
Arm/Group | BIAsp 50 | BHI 50
Serious Adverse Events (participants affected / at risk) | 1/155 | 1/158
Other Adverse Events (participants affected / at risk) | 8/155 | 2/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 50 (N=155) | BHI 50 (N=158)
Small intestinal haemorrhage (General disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 50 (N=155) | BHI 50 (N=158)
Hyperlipidaemia (Metabolism and nutrition disorders) | 8 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship of publications should be in accordance with the Uniform Requirements of the International Committee of Medical Journal Editors. The Investigators offered authorship will be asked to comment and approve the publication. No permission to publish will be granted to any clinical research organization involved in the trial described in trial protocol.